CLINICAL TRIAL: NCT02296710
Title: Echocardiographic Parameter and Sleep Apnea Changes After Mitral Valve Surgery
Acronym: MitralHDZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zisis Dimitriadis (Other)
Responsible Party: Sponsor-Investigator, Zisis Dimitriadis, Resident - Cardiologist, Heart and Diabetes Center North-Rhine Westfalia
Organization: Heart and Diabetes Center North-Rhine Westfalia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HDZNRW_KA_003_ZD
Record Dates: First submitted 2014-10-30; First posted 2014-11-20 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Sleep Apnea
Keywords: mitral valve; valve surgery; echocardiography
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Echocardiographic and sleep apnea test (Experimental): Echocardiographic Evaluation of systolic and diastolic function of both ventricles and evaluation of apnea-hypopnea index and type of apnea
  Interventions: Procedure: Echocardiographic and sleep apnea test

INTERVENTIONS:
Procedure: Echocardiographic and sleep apnea test — Echocardiographic evaluation (Vivid 7, GE) of systolic and diastolic function of both ventricles as well as evaluation of apnea-hypopnea index and type of apnea (ApneaLink®)

SUMMARY:
The investigators evaluate the changes of echocardiographic and sleep apnea parameters after mitral valve surgery. The patients undergo echocardiographic and sleep apnea control before surgery. After a period of 3-5 months, they undergo a second echocardiographic and sleep apnea control and the results are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* mitral valve defect
* NYHA II-IV
* no additional cardiac surgical procedure

Exclusion Criteria:

* Pregnancy
* lung disease
* regular follow-up in the study Center in the first 6 months after surgery not guaranteed
* congenital heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2014-08; Primary Completion 2015-05 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Changes of left ventricular systolic function | 1-4 weeks before and 3 months after surgery
Changes of apnea-hypopnea index | 1-4 weeks before and 3 months after surgery
Changes of global longitudinal strain | 1-4 weeks before and 3 months after surgery
Changes of right ventricular systolic function | 1-4 weeks before and 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zisis Dimitriadis, MD, Principal Investigator — Clinic for Cardiology, Heart and Diabetes Center North Rhine-Westphalia
Locations (1):
- Heart and Diabetes Center North Rhine-Westphalia, Bad Oeynhausen, Germany